CLINICAL TRIAL: NCT07302035
Title: A Phase Ia Single-Center, Randomized, Double-Blind, Placebo-Controlled, Safety, Tolerability, and Pharmacokinetic Trial of GenSci142 Administered in Single Ascending Doses in Healthy Chinese Women
Brief Title: A First-in-Human Safety and Pharmacokinetic Trial of GenSci142 Administered as Single Ascending Doses in Healthy Chinese Women
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: Huashan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GenSci142-101
Record Dates: First submitted 2025-11-27; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Bacterial Vaginosis
Keywords: Bacterial Infections; Vaginitis; Vaginal Diseases; Genital Diseases, Female; Female Urogenital Diseases; Gardnerella spp.; Gardnerella vaginalis; GenSci142
MeSH Terms: conditions — Vaginosis, Bacterial; Bacterial Infections; Vaginitis; Vaginal Diseases; Genital Diseases, Female; Female Urogenital Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GenSci142 (Experimental): Single ascending dose levels，All subjects administered Single dose，Dose 1, Dose 2, Dose 3
  Interventions: Drug: GenSci142
- Placebo (Placebo Comparator): All subjects administered Single dose
  Interventions: Drug: Placebo GenSci142

INTERVENTIONS:
Drug: GenSci142 — Vaginal insert
  Arms: GenSci142
Drug: Placebo GenSci142 — Vaginal insert
  Arms: Placebo

SUMMARY:
This is a Phase Ia single-center, randomized, double-blind, placebo-controlled study to assess the safety, tolerability, Pharmacokinetic of GenSci142 in Chinese healthy women.

DETAILED DESCRIPTION:
This is a Phase 1a trial including single ascending dose levels and will assess the safety and tolerability of GenSci142 and describe the incidence of adverse events (AEs) for participants randomized at a ratio of 4:1 to GenSci142 or placebo within each cohort. Participants will receive one single dose of study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women of childbearing potential aged 18-55 years (inclusive) at the time of signing the Informed Consent Form (ICF);
* Sexually active and willing to undergo vaginal administration of the study product；participants must agree to avoid the use of other intravaginal products (e.g., contraception ointments, gels, foams, sponges, lubricants, irrigation solutions, tampons, etc.) throughout the trial;
* During the screening period, there are no clinically significant abnormalities in medical history, vital signs, physical examination, gynecological examination, laboratory test (hematology, routine urinalysis, clinical chemistry, coagulation function, vaginal microbiome test) and 12-lead ECG, or any out-of-range laboratory values or other findings must be assessed by the investigator as not clinically significant;

Exclusion Criteria:

* Those experiencing stinging or burning sensation, hemorrhage, pruritus, erythema, edema, or increased discharge due to previous or current use of vaginal preparations, or those with any factors that possibly have an impact on evaluation of administration site irritation, or those with other factors that may have an impact on vaginal administration, such as genital malformation;
* Serious infections, chronic infections, opportunistic infections, etc. within 3 months prior to screening, and infections treated with systemic antimicrobial drugs (including but not limited to viruses, bacteria, fungi, and parasitic infections) within 4 weeks prior to randomization;
* Surgical history: a. vaginal, pelvic or cervical surgery within 90 days prior to screening or planning to undergo surgery during the study; b. hysterectomy; c. other major surgery within 30 days prior to screening or planning to undergo other surgeries during the study;

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with adverse events (AEs) with onset after dose and until 15 days post-dose | from first dose of study treatment up to 15 days post-dose
  In participants who have received at least one dose of GenSci142 or placebo. For each dose level cohort of GenSci142 and for the placebo group.

SECONDARY OUTCOMES:
Serum concentration of GenSci142 (ng/mL) | Day1-Day3
  Concentrations of GenSci142 in serum samples at different time points are measured. Serum concentrations at different time points will be listed and summarized by descriptive statistics.
Maximum serum concentration (Cmax, ng/mL) | Day1-Day3
  PK parameters will be analyzed by non-compartmental analysis with WinNonlin® version 8.3 or above.
Time to maximum serum concentration (Tmax, h) | Day1-Day3
  PK parameters will be analyzed by non-compartmental analysis with WinNonlin® version 8.3 or above.
Area under the concentration-time curve from the time zero to last measurable concentration (AUC0-t, h*ng/mL) | Day1-Day3
  PK parameters will be analyzed by non-compartmental analysis with WinNonlin® version 8.3 or above.
Area under concentration-time from time zero to infinity (AUC0-inf, h*ng/mL) | Day1-Day3
  PK parameters will be analyzed by non-compartmental analysis with WinNonlin® version 8.3 or above.
Terminal half-life (t1/2, h) | Day1-Day3
  PK parameters will be analyzed by non-compartmental analysis with WinNonlin® version 8.3 or above.
Apparent clearance (CL/F, mL/h) | Day1-Day3
  PK parameters will be analyzed by non-compartmental analysis with WinNonlin® version 8.3 or above.
Apparent volume of distribution (Vd/F, mL) | Day1-Day3
  PK parameters will be analyzed by non-compartmental analysis with WinNonlin® version 8.3 or above.
Anti-drug antibody (ADA) prevalence (%) or change of binding titers against GenSci142 in blood before administration and at the follow-up visit | Day1-Day15
  For each dose level.

CONTACTS AND LOCATIONS:
Overall Officials: Jing ZHANG, Doctor, Study Chair — Huashan Hospital
Locations (1):
- Huashan Hospital Fudan University, Shanghai, Shanghai Municipality, China